CLINICAL TRIAL: NCT07132164
Title: Justification of the Initial Diagnosis and Evaluation of the Overall Evolution of a Cohort of Recent Polymyalgia Rheumatica
Brief Title: Justification of the Initial Diagnosis and Evaluation of the Overall Evolution of a Cohort of Recent Polymyalgia Rheumatica (JADORE)
Acronym: JADORE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0391; 2024-A00863-44 (Other: IDRCB)
Record Dates: First submitted 2025-07-08; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Polymyalgia Rheumatica; Inflammatory Rheumatism
Keywords: polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica; Rheumatic Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At inclusion, patients will benefit from blood testing for biobank establishment, and stool sample collection for gut microbiota analysis will be organized depending on the center. The 12-month visit (M12) will also include an additional blood sample collection as part of the biobank, as well as stool sample collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biological sample collection: Biobank establishment and stool sample collection for gut microbiota analysis
  Interventions: Other: biobank sample collection

INTERVENTIONS:
Other: biobank sample collection — At inclusion, patients will benefit from blood testing for biobank establishment, and stool sample collection for gut microbiota analysis will be organized depending on the center.
  The 12-month visit (M12) will also include an additional blood sample collection as part of the biobank, as well as stool sample collection

SUMMARY:
Pseudo-rheumatoid arthritis (PRA) is a common inflammatory rheumatic disease of the elderly, characterized by inflammatory shoulder and/or hip pain. Its routine diagnosis is based on a number of clinical criteria, the presence of a biological inflammatory syndrome and the elimination of the main differential diagnoses. It is sometimes referred to as PPR syndrome, since around 25% of initial diagnoses are not confirmed at one year's follow-up (PPR syndrome revealing rheumatoid arthritis, microcrystalline rheumatism, etc.). Diagnosis may be facilitated by ultrasound scans of the shoulders and hips, which may show characteristic inflammatory lesions, or by PET scans when there is a marked deterioration in general condition or other clinical atypia. PPR may be associated at the outset, or it may evolve into the rarer vasculitis of the elderly, giant cell arteritis (GCA), a condition that can lead to severe and irreversible neurological vascular damage if not treated early.

Prolonged, moderate-dose corticosteroid therapy is the cornerstone of PPR treatment, although new treatments are in the process of obtaining marketing authorization to enable cortisone sparing. Anti-IL-6 agents, and in particular Tocilizumab, have demonstrated their efficacy in recent cortico-dependent PPR, Sarilumab has obtained marketing authorization for cortico-dependent PPR in the USA in 2023, and other therapeutic classes are currently being evaluated in this situation. Recommendations, including those of ACR/EULAR in 2015, advise a strategy of initiating corticosteroid therapy at a moderate dose, with a dosage of between 12.5 and 25 mg prednisone equivalent per day, and gradually tapering off with the aim of reaching a dosage of 10 mg prednisone equivalent per day at week 8, to achieve complete weaning at 12 months. However, on the one hand, these recommendations are not based on clinical trials and, on the other, the main comorbidities associated with PPR are related to this long-term corticosteroid therapy. Lastly, we know that around 50% of patients do not follow this tapering-off protocol, with either relapses (estimated at 50% during tapering) or the impossibility for around 25% of patients to stop corticosteroid therapy. However, there are currently no predictive factors for the evolution of PPR.

PPR activity can be measured either using a validated score, the DAS-PPR, or according to the opinion of the rheumatologist. Good progression of rheumatoid arthritis is characterized by a low activity score (DAS-PPR<10) and, wherever possible, discontinuation of treatment within one year, as recommended by international experts.

The main objective of this cohort is therefore to evaluate the percentage of patients with low-activity PPR (DAS-PPR<10) and no treatment at 12 months.

Secondary objectives will concern the initial phenotypic and evolutionary description of PPR (complete initial phenotypic characteristics, including some exploratory ones (imaging, biology, immunology, genetics, microbiota, avatars). The evolution of the disease, with the percentage of relapses during the decline or distant relapses, percentage of association with ACG, mortality rate, as well as the prognostic factors of these different evolutionary forms. A description of the disease-modifying treatments used (corticosteroid therapy and its decline, other immunomodulators), as well as a record of the complications presented by patients (development of ACG, corticosteroid toxicity, sarcopenia, osteoporosis fractures, diverticular perforation). Finally, many pathologies can clinically and biologically mimic PPR, leading to erroneous prescriptions of glucocorticoids for prolonged periods, and sometimes a delay in the diagnosis of serious conditions. These classic differential diagnoses will be investigated according to the clinical context and the clinician's judgement, and the diagnostic value of tests such as joint ultrasound, PET scans and biomarkers can be assessed.

With regard to patient follow-up, if an alternative diagnosis is identified immediately after the completion of additional examinations, the patient is no longer followed up in the study, and the alternative diagnosis is noted by the investigator. For patients for whom the investigator's conviction concerning the diagnosis of PPR remains above 50%, as at inclusion, follow-up in the study is continued. At one year's follow-up, if an alternative diagnosis has been made, this is collected and the patient is no longer followed up in the cohort. Follow-up for other patients then continues for 5 years. Deterministic matching to the SNDS will be performed for each patient included.

To date, there is no French prospective cohort dedicated to the follow-up of patients with a recent form of PPR, as has been done for rheumatoid arthritis, spondyloarthritis and psoriatic arthritis. The creation of such a cohort will improve our knowledge of this pathology, in terms of both pathophysiology and routine management.

DETAILED DESCRIPTION:
Participation in the study will be offered to all patients meeting the inclusion and non-inclusion criteria. Patients will be given sufficient time to reflect before confirming their participation in the study (the usual delay in obtaining the results of the initial pathology assessment before starting prolonged corticosteroid therapy means that this delay will in practice be several days in all cases). All study assessments will be carried out at visits corresponding to these patients' routine care (M0 inclusion), M3, M6, M12, M24, M36, M48 and M60. Two additional teleconsultation visits at M18 and M30 may be carried out to record major follow-up events (current treatments and dose, disease activity, treatment complications, occurrence of ACG). Patients will also be assessed at the time of their first relapse, if applicable.

At the inclusion visit, data will be collected on the complementary examinations usually carried out as part of the initial PPR work-up: standard biological work-up, immune work-up, chest X-ray, shoulder and pelvis X-rays, and bone densitometry. Data concerning the performance of a PET scan or MRI of the shoulders will also be collected. Patients will have a blood test to build up the biocollection, and a stool sample (depending on the center) will be collected to study intestinal microbiota. Patients will receive ultrasound scans of the hips and shoulders as part of their routine care. Doppler ultrasound of the supra-aortic trunks will be performed (at extra cost). Quality-of-life questionnaires will be completed. Sarcopenia will be assessed using the SARC-F self-questionnaire, SPPB muscle performance measurement, Handgrip test muscle strength and frailty syndrome.

Patients for whom the clinician's conviction is less than 50% after the initial complementary assessment will not be followed up in the cohort. At one year's follow-up, if the clinician's conviction remains > 50%, patients will be followed up in the study. For the others, follow-up will be stopped.

Follow-up visits and the additional visit at the time of the first relapse will include the collection of clinical, biological and imaging data corresponding to routine care, as well as the administration of quality-of-life questionnaires. The visit at M12 will also include additional blood collection as part of the biocollection and the collection of a stool sample.

Throughout the study, the daily and cumulative dosage of glucocorticoids and immunosuppressants actually received by patients will be collected via a paper logbook or a dedicated application (internet/redcap or Smartphone).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 50, with no upper age limit
* Inflammatory shoulder +/- hip pain
* Abnormal CRP (≥10mg/L)
* Patients for whom the referring rheumatologist accepts the diagnosis of PPR after carrying out the assessment corresponding to his or her current practice
* Patients for whom the referring rheumatologist has indicated that corticosteroid therapy should be started in the strict context of PPR or as background treatment for PPR.
* Symptoms have progressed for 24 weeks or less

Exclusion Criteria:

* Presence, at the time of diagnosis, of symptoms and/or signs suggesting a diagnosis of associated giant cell arteritis
* Immuno-induced PPR
* Patients receiving immunosuppressive treatment with methotrexate or immunotherapy targeting interleukin-6 at inclusion.
* Patients who have received corticosteroid therapy for more than 30 days or a cumulative dose of more than 500 mg of Prednisone equivalent in the month preceding the screening visit.
* Patients with another chronic condition requiring long-term corticosteroid therapy or repeated courses of corticosteroids.
* Patients not affiliated to a social security scheme
* Patients unable to consent or unable or unwilling to complete their corticosteroid dose monitoring record.
* Pregnancy
* Patients under guardianship, curatorship or safeguard of justice

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients agreeing to take part in the study and meeting the inclusion and non-inclusion criteria will be referred to the nearest rheumatology department participating in the study
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of DAS-PPR (Disease Activity Score) | 12 months
Number of participants with no PPR-related treatment for at least 2 weeks | 12 months

SECONDARY OUTCOMES:
Number of patients with a Diagnosis of PPR maintained | Months 12, 24, 36, 48, 60, First relapse within 5 years of follow-up
  Medical reassessment of patients for diagnostic reassessment
Classification criteria ACR/EULAR (American College of Rheumatology/European Alliance of associations for rheumatology) 2012 | Inclusion
Shoulder and hip ultrasound score | Inclusion
Measurement of the Leuven score | Inclusion
Definitive diagnosis of PRA according to the expert clinican | Month 24
Characteristics of clinical PRA (collection of affected joints) | Inclusion
Characteristics of clinical PRA (CRP level) | Inclusion
Alternative diagnosis retained by the expert clinician: microcrystalline inflammatory rheumatism; other chronic inflammatory rheumatic diseases ; paraneoplastic rheumatism | Inclusion, Month 12, 24, 36, 48 and 60
Measurement of DAS-PPR (Disease Activity Score) | Inclusion, Month 3, 6, 12, 24, 36, 48, 60, First relapse within 5 years of follow-up
Remission: DAS-PPR < 10, no corticosteroids, and no immunomodulatory treatments | Inclusion, Month 3, 6, 12, 24, 36, 48, 60
Relapse: Reinitiation of corticosteroids or immunomodulatory therapy | Inclusion, Month 3, 6, 12, 24, 36, 48, 60
Number of patient with a Diagnosis of Giant Cell Arthritis during the follow-up of the study | Month 3, 6, 12, 24, 36, 48, 60, First relapse within 5 years of follow-up
Measurement of SF36 | Inclusion, Month 3, 6, 12, 24, 36, 48, 60, First relapse within 5 years of follow-up
Measurement of EQ-5D | Inclusion, Month 3, 6, 12, 24, 36, 48, 60, First relapse within 5 years of follow-up
Death occurence | Month 3, 6, 12, 24, 36, 48, 60
Adverse events characteristic of PPR | Month 3, 6, 12, 24, 36, 48, 60, First Relapse within 5 years of follow-up
Dosage of glucocorticoids | Inclusion, Month 3, 6, 12, 24, 36, 48, 60, First relapse within 5 years of follow-up
Measurement of Glucocorticoid toxicity with the Glucocorticoid toxicity index, gti score | Inclusion, Month 3, 6, 12, 24, 36, 48, 60, First relapse within 5 years of follow-up
Change in lipid parameters | Inclusion, Month 12
Change in glycemic parameters | Inclusion, Month 12
Measurement of bone densitometry parameters | Inclusion, Month 12
Number of Fracture event | Month 3, 6, 12, 24, 36, 48, 60
Number of falls self-reported by patients | Month 12, 24, 26, 48, 60
Cumulative dose of corticosteroids received by the patient since inclusion | Month 12, 24, 36, 48, 60
Relapse rate after stopping immunomodulators | Month 3, 6, 12, 24, 36, 48, 60, First relapse within 5 years of follow-up
SARC-F self-questionnaire | Inclusion, M12, M36, M60, First relapse within 5 years of follow-up
Handgrip measure with handgrip test | Inclusion, M12, M36, M60, First relapse within 5 years of follow-up
Short Physical Performance Battery | Inclusion, M12, M36, M60, First relapse within 5 years of follow-up
Occurence of Gastrointestinal perforations | Inclusion, M12, M36, M60, First relapse within 5 years of follow-up
Major adverse cardiovascular events | Inclusion, M12, M36, M60, First relapse within 5 years of follow-up
Measuring the Groll index | Inclusion, Month 6, 12, 24, 36, 48, 60
Measurement of the Fragility Score (FRIED) | Inclusion, Month 12, 36, 60, First relapse within 5 years of follow-up
Serum and transcriptomic biomarkers | Inclusion

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - CHU Rouen, Rouen, Rouen
  - Besançon-CIC, Besançon
  - CHU Besançon, Besançon
  - CHU de Bordeaux Pellegrin, Bordeaux
  - CH Boulogne/mer, Boulogne-sur-Mer
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - Clinique de l'Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH Dax, Dax
  - CHU de Dijon, Dijon
  - CH La Roche s/ Yon, La Roche-sur-Yon
  - APHP - Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHU de Lille, Lille
  - Institut catholique de Lille, Lomme
  - CHU Marseille AP-HM, Marseille
  - CH Le Havre, Montivilliers
  - CHU de Montpellier, Montpellier
  - CH Morlaix, Morlaix
  - CHU de Nice, Nice
  - AP-HP La Pitié-Salpétrière, Paris
  - AP-HP Cochin, Paris
  - AP-HP Bichat, Paris
  - Hopital NOVO - Site Pontoise, Pontoise
  - CHU Saint-Etienne, Saint-Priest-en-Jarez
  - CHU Strasbourg, Strasbourg
  - Clinique Ambroise Paré-Toulouse, Toulouse
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided